CLINICAL TRIAL: NCT06437015
Title: Comparison of CIMT vs Mirror Therapy Effect in Infarcted CVA Patients for Improving Hand Functions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/720
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Infected Joint
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-Induced Movement Therapy (Experimental)
  Interventions: Diagnostic Test: Constraint-Induced Movement Therapy
- Mirror Therapy (Active Comparator)
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Diagnostic Test: Constraint-Induced Movement Therapy — patient's unaffected hand is tied with a triangular bandage or splint and the patient asks to perform the exercise through the affected hand. for up to 6 hours a day for 5days week /4 weeks and the patient nonparetic arm restrained from the use by having the patient placing a mitt on the hand or a sling on the unaffected hand, forcing the use of the affected limb to promote purposeful movements when performing functional tasks.
  Arms: Constraint-Induced Movement Therapy
Other: Mirror Therapy — In this group training was given for 45min a day for 5 days a week for 4 weeks. Mirror box which was of 18×24inch [was placed on the learning table and exercises were carried out by the patient looking into the mirror where an unaffected limb is placed in front of the mirror, through looking into the mirror patient assumes the reflection of the unaffected limb as the paretic limb. Exercises performed were hand opening and closing, wrist extension and flexion, squeezing, opposition, the calculation
  Arms: Mirror Therapy

SUMMARY:
CIMT vs Mirror therapy for improving hand function in infarcted CVA patients. Randomized clinical trial study design will be followed. Data will be collected from following centers: Minhaj Physiotherapy Centre, Home visits, Sughra sidiq trust hospital, Ibad hospital Samundri. Probability Random Sampling is used.

ELIGIBILITY:
Inclusion Criteria:

* Infarcted CVA patients
* Patients with hand improvement needed
* Patients in recovery stage of stroke from 2 months to 1 year
* Patients who can participate in 45 mins of session

Exclusion Criteria:

* Patients with hand function disturbed due to any other reason except infarcted CVA, - - - Patients with shoulder subluxation and upper limb contractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment (FMA) | 12 Months
  it is a stroke-specific, performance-based impairment index.Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully
The Chedoke Arm and Hand Activity Inventory (CAHAI) | 12 months
  It is used to assess functional ability of the paretic arm and hand. This test consists of 13 functional tasks: open a jar of coffee, draw a line with a ruler, put toothpaste on a toothbrush, cut medium consistency putty,pour a glass of water wring out a washcloth,clean a pair of eyeglasses,zip up a zipper,botton up 5 buttons,dry back with a towel,place a container on a table and carry a bag up the stairs.

CONTACTS AND LOCATIONS:
Locations (1):
- Minhaj Physiotherapy, opp Shalimar Hospital , Shalimar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No